CLINICAL TRIAL: NCT00839579
Title: How Little Pain for Cardiac Gain? A Pilot Study
Brief Title: Cardiovascular Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1x4min interval
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: slightly overweight; males 35-45 years
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4x4min (Experimental): 4x4minutes interval group
  Interventions: Other: 1x4 min interval
- 1x4min (Experimental)
  Interventions: Other: 1x4 min interval

INTERVENTIONS:
Other: 1x4 min interval — Aerobic interval training

SUMMARY:
Exercise training is proved to protect against premature cardiovascular mortality. Additionally there is evidence that relatively high exercise intensity may be an important factor for improving aerobic capacity and endothelial function in patients with post-infarction heart failure, metabolic syndrome, coronary artery disease, as well as in overweight and obese individuals.

The aim of this study is to investigate the amount of high-intensity exercise needed to improve aerobic capacity and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-30
* Males, 35-45 years
* Healthy

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption and endothelial function | baseline and 12 weeks followup

CONTACTS AND LOCATIONS:
Overall Officials: Arnt E Tjønna, PhD, Study Chair — Norwegian University of Science and Technology; Ulrik Wisløff, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Tjonna AE, Leinan IM, Bartnes AT, Jenssen BM, Gibala MJ, Winett RA, Wisloff U. Low- and high-volume of intensive endurance training significantly improves maximal oxygen uptake after 10-weeks of training in healthy men. PLoS One. 2013 May 29;8(5):e65382. doi: 10.1371/journal.pone.0065382. Print 2013. PMID 23734250